CLINICAL TRIAL: NCT07407387
Title: Appropriateness of Medication Prescribing in Nursing Homes: A Pre-Post Study to Evaluate the Effectiveness of a Clinical Pharmacology Team-Led, Digitally Supported, Inter-Professional Collaboration
Brief Title: Ensuring Clinical Appropriateness and Safety of Pharmacological Therapies in Nursing Home Residents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lugano Istituti Sociali (Other)
Collaborators: Ente Ospedaliero Cantonale, Ticino, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISFSI_LIS_2025
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Inappropriate Prescribing

STUDY DESIGN:
Intervention Model Description: Pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Appropriateness of medication prescribing (Experimental): Confirmatory, single-arm, non-randomized, pre-post study conducted in the geriatric clinical setting of seven nursing homes located in Southern Switzerland, coordinated by Lugano Istituti Sociali (LIS), in collaboration with the Institute of Pharmacological Sciences of Southern Switzerland and the Clinical Trial Unit of the Ente Ospedaliero Cantonale (ISFSI-EOC and CTU-EOC).
  Each resident will serve as their own control, with outcomes measured over a 3-month pre-intervention period and a 3-month post-intervention period. The intervention, lasting approximately 3 months, includes individualized medication review by clinical pharmacologists, face-to-face feedback and tailored educational sessions for nursing home healthcare professionals responsible for managing residents' medications.
  Interventions: Procedure: Multi-Component Intervention on Medication Prescribing

INTERVENTIONS:
Procedure: Multi-Component Intervention on Medication Prescribing — The study intervention is a multi-component procedure led by a team of clinical pharmacologists to improve medication prescribing among nursing home residents. It includes: 1) individualized medication review with a comprehensive review of each resident's medications, digitally supported; the assessment of medication prescribing appropriateness using the Medication Appropriateness Index (MAI), the identification of key indicators of inappropriate prescribing and the assessment of resident-centred clinical outcomes; 2) face-to-face feedback with nursing home healthcare professionals responsible for managing residents' medications to discuss recommended adjustments for each resident, fostering inter-professional collaboration; 3) tailored educational sessions to nursing home healthcare professionals responsible for managing residents' medications, addressing common prescribing issues identified during medication review. No drugs or medical devices will be used during this procedure.

SUMMARY:
The goal of this clinical study is to evaluate whether a structured, clinical pharmacology team-led medication review improves the appropriateness and safety of medication prescribing in elderly nursing home (NH) residents. The study will also assess the impact of the intervention on indicators of inappropriate prescribing and resident-centred clinical outcomes. The main questions the study aims to answer are: 1) Does a structured, digitally supported, medication review led by clinical pharmacologists reduce inappropriate medication prescribing, as measured by the Medication Appropriateness Index (MAI), in elderly NH residents? 2) Does the intervention reduce indicators of inappropriate prescribing, including potentially inappropriate prescriptions, therapeutic duplicates, drug-drug interactions and anticholinergic burden? 3) Does the intervention improve resident-centred clinical outcomes, such as falls, fractures, delirium, hyper-sedation, emergency department visits and hospitalizations? This is a single-arm, non-randomized, pre-post study conducted in seven NHs in Southern Switzerland. Each resident will serve as their own control, with outcomes compared between a 3-month pre-intervention period and a 3-month post-intervention period.

The intervention consists of: 1) An individualized, digitally supported, medication review conducted by the team of clinical pharmacologists; 2) Face-to-face feedback to NH healthcare professionals responsible for managing residents' medications; 3) Tailored educational sessions addressing common prescribing issues identified during the medication review.

Participants will: be aged 65 years or older and reside in participating NHs; have their routinely collected clinical and medication data assessed during a 3-month pre-intervention period; receive the intervention integrated into routine care, with any medication changes implemented by treating clinicians.

The study is low-risk, non-invasive, and embedded in routine NH care. The results will provide evidence on the clinical effectiveness of integrating clinical pharmacology expertise into inter-professional medication management in Swiss NHs.

ELIGIBILITY:
Inclusion Criteria:

* Expected to remain in the nursing home for the duration of the study
* Able to provide informed consent or having a legally authorized representative able to provide consent if the resident lacks capacity

Exclusion Criteria:

* Residents in their probable last hours or days of life
* Residents with moderate to severe cognitive impairment (Cognitive Performance Scale, CPS, score >4
* Residents housed in assisted nursing home wards, including those requiring palliative care (either in dedicated palliative units or receiving palliative care in general wards), those in the hemodialysis unit, and those with severe obesity (body mass index >=40kg/m2)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Medication Appropriateness Index (MAI) | Pre-intervention (day 1) and post-intervention (day 180), for comparison
  Reduction in the total MAI score per resident between pre-intervention (day 1) and post-intervention (day 180) periods. The MAI is calculated at the medication level for each long-term in-use medication (>=3 months, excluding as needed medications), using a modified 10-item MAI scoring system. Each medication is scored from 0 to 17 (higher score=greater inappropriateness). A resident-level MAI is calculated by summing the MAI scores of all eligible medications.

SECONDARY OUTCOMES:
Indicators of inappropriate prescribing | Pre-intervention (day 1) and post-intervention (day 180), for comparison
  Frequency of indicators of inappropriate prescribing, including potentially inappropriate prescriptions (PIPs), therapeutic duplicates (TDs), drug-drug interactions (DDIs), and anticholinergic burden (ACB).
  These indicators will be determined for each participant based on the individual medication list. Specifically, PIPs will be identified according to the American Geriatrics Society Updated Beers Criteria for Potentially Inappropriate Medication Use in Older Adults (2023); TDs will be defined as the concurrent prescription of two or more drugs within the same Anatomical Therapeutic Chemical (ATC) subgroup at the fourth level; DDIs will be assessed by clinical pharmacologists through consultation of Lexicomp (external drug interaction database); and ACB will be evaluated by clinical clinical pharmacologists according to the ACB scale 2012.
Resident-centred clinical outcomes | Pre-intervention (day 1) and post-intervention (day 180), for comparison
  Frequency of falls, fractures, delirium, hyper-sedation, drug-related emergency department visits and hospitalizations.
  The occurrence of the specified outcomes will be ascertained through extraction of data from the electronic health records of nursing home residents, where such information is routinely recorded as part of standard clinical documentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Pharmacological Science of Southern Switzerland, Ente Ospedaliero Cantonale, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No